CLINICAL TRIAL: NCT03005366
Title: Randomized Clinical Trial to Study Pharmacological Cardioversion of Paroxysmal Atrial Fibrillation by Vernakalant and Flecainide
Brief Title: Predictive Factors to Effectively Terminate Paroxysmal Atrial Fibrillation by Blocking Atrial Selective Ionic Currents
Acronym: SELECTCARFAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: David Filgueiras-Rama (Other)
Collaborators: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor-Investigator, David Filgueiras-Rama, MD PhD, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELECTI-CARFAP
Record Dates: First submitted 2016-12-05; First posted 2016-12-29 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial fibrillation; vernakalant; flecainide; cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — vernakalant; Flecainide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flecainide (Active Comparator): Conventional cardioversion group using intravenous flecainide.
  Interventions: Drug: Flecainide
- Vernakalant (Active Comparator): Atria-preferential and atrial-specific blockade group using intravenous vernakalant.
  Interventions: Drug: Vernakalant

INTERVENTIONS:
Drug: Vernakalant — Initial infusion: 3 mg/kg intravenously over a 10 minute period. For patients weighing ≥ 113 kg, the maximum initial dose will be 339 mg. If conversion to sinus rhythm does not occur within 15 minutes after the end of the initial infusion, a second 10 minute infusion of 2 mg/kg will be administered. For patients weighing ≥ 113 kg, the maximum second infusion will be 226 mg.
  Other Names: BRINAVESS
  Arms: Vernakalant
Drug: Flecainide — 2 mg /kg (max 150 mg) intravenously over 10 minutes.
  Other Names: APOCARD
  Arms: Flecainide

SUMMARY:
* The main objective of this project is to study the efficacy and the mechanistic value of blocking both atrial specific and atria-preferential dynamics of ionic currents to terminate paroxysmal atrial fibrillation (AF).
* The hypothesis is that a drug blocking atrial specific and atria-preferential dynamics of ionic currents (IK,ACh - acetylcholine sensitive K+ current - and INa - inward sodium current - , respectively) will be more effective to terminate paroxysmal AF episodes with fast atrial activation rates, than a classical INa blocker, which will be more effective to terminate AF episodes with slower activation rates.
* The investigators will include patients without structural heart disease and short-lasting AF episodes (<48 h.). Double blind and single center study, in which patients will be randomly assigned to a cardioversion group using intravenous flecainide or to an atria-preferential and atrial-specific blockade group using intravenous vernakalant. Patients will be routinely monitored in the electrophysiology room to acquire both 12-lead digitized ECG signals and non-invasive body surface potential mapping. Atrial signals will be extracted from both the multisite body surface and ECG recordings to obtain temporal and spectral parameters, and measure organization and atrial rate in both groups. The results obtained in the clinical setting will be studied in mathematical models to understand their capability to terminate paroxysmal AF. The project expects to provide consistent, reliable and reproducible parameters that will assist clinicians to know what type of paroxysmal AF episodes will be more suitable to effectively terminate, upon administration of drugs with an atrial specific and atria-preferential profile.

DETAILED DESCRIPTION:
* Background: Different research strategies aim at understanding the mechanisms underlying the maintenance of atrial fibrillation (AF), while preventing ventricular pro-arrhythmia related to the use of anti-arrhythmic drugs to restore sinus rhythm. Such aims might be achieved by drugs that effectively terminate reentrant sources identified during AF, along with an atrial specific and atria-preferential blockade of ionic currents. The latter may be especially relevant in paroxysmal AF episodes with fast atrial activation rates, in which INa and IK,ACh are involved in the maintenance of fast atrial reentrant sources underlying AF.
* Objective: The main objective of this project is to study the efficacy and the mechanistic value of blocking both atrial specific and atria-preferential dynamics of ionic currents to terminate paroxysmal AF.
* The hypothesis is that a drug blocking atrial specific and atria-preferential dynamics of ionic currents (IK,ACh and INa, respectively) will be more effective to terminate paroxysmal AF episodes with fast atrial activation rates, than a classical INa blocker, which will be more effective to terminate AF episodes with slower activation rates.
* Design: Double blind and single center study, in which patients will be randomly assigned to a cardioversion group using intravenous flecainide or to an atria-preferential and atrial-specific blockade group using intravenous vernakalant. Patients will be routinely monitored in the electrophysiology room for 90 minutes upon drug administration to acquire both 12-lead digitized ECG signals and non-invasive body surface potential mapping. Body surface recordings and conventional ECG signals will be exported to obtain temporal and spectral parameters of atrial activity during AF, and measure organization and atrial rate in both groups of patients undergoing pharmacological cardioversion. The success rate of cardioversion obtained in both groups will be correlated with the patterns of activation and spectral parameters obtained from the body surface, which will provide what type of paroxysmal AF episodes are suitable to terminate upon administration of anti-arrhythmic drugs with an atrial specific and atria-preferential profile.

Electrical cardioversion will be performed in subjects with unsuccessful pharmacological cardioversion within the first 24 h. after vernakalant or flecainide administration.

The results obtained in the clinical setting will be studied in realistic mathematical models to further understand the capability of both drugs to terminate paroxysmal AF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 20 and ≤65 year-olds.
2. Patients with paroxysmal AF lasting <48 hours, in whom pharmacological cardioversion may be indicated.
3. Hemodynamically stable patients (systolic blood pressure > 100 mm Hg and < 160 mm Hg. Diastolic blood pressure <95 mm Hg).
4. Weight of 45-136 kg .
5. Appropriate anticoagulation therapy according to the clinical practice guidelines of the European Society of Cardiology in paroxysmal AF episodes lasting < 48 hours.
6. Signed informed consent.

Exclusion Criteria:

1. Corrected QT interval> 440 milliseconds, long QT family or history of 'Torsades de Pointes' syndrome.
2. Symptomatic bradycardia or ventricular rate <50 bpm without a pacemaker, or QRS interval> 140 milliseconds.
3. Patients with heart failure regardless of the classification of the New York Heart Association (NYHA).
4. Second or third degree atrioventricular block, or right bundle branch block associated with partial left bundle branch block (bifascicular block).
5. Cardiogenic or septic shock, chronic myocardial infarction, acute coronary syndrome, or heart surgery in the previous 30 days before inclusion.
6. Valvular stenosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis.
7. Previous unsuccessful electrical cardioversion or longstanding atrial fibrillation (no attempt to convert to sinus rhythm).
8. Treatment with other investigational drug within 60 days before enrollment.
9. Previous treatment with vernakalant.
10. Secondary causes of atrial fibrillation, hyperthyroidism, uncorrected electrolyte imbalance, or digoxin toxicity.
11. IV / oral treatment with Class I or III antiarrhythmics (except amiodarone) in the previous 48 hours.
12. Renal failure with glomerular filtration rate <35 ml / min.
13. Intravenous / oral amiodarone within the previous 3 months.
14. Pregnant or nursing women.
15. Intolerance or allergy to any of the two drugs being studied.
16. Refusal to sign the informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Electrocardiographic-based spectral parameters of atrial fibrillatory activity (Dominant frequency) associated with successful or unsuccessful cardioversion in both groups of patients. | 18 months
  The investigators will quantify the difference in baseline dominant frequency values (Hz) of atrial fibrillatory activity between patients with successful cardioversion in the vernakalant and flecainide groups.
  The investigators will also quantify the difference in baseline dominant frequency values (Hz) of atrial fibrillatory activity between patients with successful and unsuccessful cardioversion within the vernakalant or flecainide group.

SECONDARY OUTCOMES:
Cardioversion success (yes/no) in patients with paroxysmal atrial fibrillation episodes lasting < 24 hours or ≥24 hours. | 18 months
  The investigators will quantify the difference in cardioversion success (yes/no) between episodes lasting < 24 hours or ≥24 hours.
Electrocardiographic-based spectral parameters of atrial fibrillatory activity (Dominant frequency) in patients with episodes lasting < 24 hours or ≥24 hours. | 18 months
  The investigators will quantify the difference in baseline dominant frequency values (Hz) of atrial fibrillatory activity between patients with episodes lasting < 24 hours or ≥24 hours.
Spectral parameters of atrial fibrillatory activity (Dominant frequency) recorded by non-invasive body surface potential mapping associated with successful or unsuccessful cardioversion in both groups of patients. | 24 months
  The investigators will quantify the difference in baseline dominant frequency values (Hz) of atrial fibrillatory activity between patients with successful cardioversion in the vernakalant and flecainide groups.
  The investigators will also quantify the difference in baseline dominant frequency values (Hz) of atrial fibrillatory activity between patients with successful and unsuccessful cardioversion within the vernakalant or flecainide group.
Effects on reentrant-based atrial fibrillation (dominant frequency decrease, rotor meandering) in 2D models of fast and low atrial activation rates under the effect of vernakalant or flecainide. | 24 months
  The investigators will quantify dominant frequency changes (Hz) and rotor meandering (mm) under the effect of vernakalant or flecainide in 2D computational models.
Atrial Fibrillation Quality of Life questionnaire (AF-QOL). | 24 months
  The Investigators will quantify the effects of atrial fibrillation on patients´ quality of life base on of the Atrial Fibrillation Quality of Life questionnaire (AF-QOL).

OTHER OUTCOMES:
Patient's perception during cardioversion. The investigators will used a custom-designed five-question questionnaire as follows: | 24 months
  i) Do you recall something from the cardioversion attempt? yes/no. ii) If (1) is yes, was it uncomfortable? yes/no. iii) Did you feel any pain during the cardioversion attempt? yes/no. iv) Please, provide an score from '0' to '10' to evaluate your general perception of the cardioversion attempt.
  v) If necessary, would you undergo another cardioversion attempt using the same strategy? yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Nicasio Pérez-Castellano, MD, PhD, Study Chair — Hospital San Carlos, Madrid; Asunción Conde, PharmD, Study Chair — Hospital San Carlos, Madrid; María-Jesús García-Torrent, PharmD, PhD, Study Chair — Hospital San Carlos, Madrid
Locations (1):
- Hospital Clínico Universitario San Carlos, Madrid, Madrid/Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kannel WB, Wolf PA, Benjamin EJ, Levy D. Prevalence, incidence, prognosis, and predisposing conditions for atrial fibrillation: population-based estimates. Am J Cardiol. 1998 Oct 16;82(8A):2N-9N. doi: 10.1016/s0002-9149(98)00583-9. PMID 9809895
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Mandapati R, Skanes A, Chen J, Berenfeld O, Jalife J. Stable microreentrant sources as a mechanism of atrial fibrillation in the isolated sheep heart. Circulation. 2000 Jan 18;101(2):194-9. doi: 10.1161/01.cir.101.2.194. PMID 10637208
- [Background] Gray RA, Jalife J, Panfilov AV, Baxter WT, Cabo C, Davidenko JM, Pertsov AM. Mechanisms of cardiac fibrillation. Science. 1995 Nov 17;270(5239):1222-3; author reply 1224-5. No abstract available. PMID 7502055
- [Background] Berenfeld O, Mandapati R, Dixit S, Skanes AC, Chen J, Mansour M, Jalife J. Spatially distributed dominant excitation frequencies reveal hidden organization in atrial fibrillation in the Langendorff-perfused sheep heart. J Cardiovasc Electrophysiol. 2000 Aug;11(8):869-79. doi: 10.1111/j.1540-8167.2000.tb00066.x. PMID 10969749
- [Background] Sanders P, Berenfeld O, Hocini M, Jais P, Vaidyanathan R, Hsu LF, Garrigue S, Takahashi Y, Rotter M, Sacher F, Scavee C, Ploutz-Snyder R, Jalife J, Haissaguerre M. Spectral analysis identifies sites of high-frequency activity maintaining atrial fibrillation in humans. Circulation. 2005 Aug 9;112(6):789-97. doi: 10.1161/CIRCULATIONAHA.104.517011. Epub 2005 Aug 1. PMID 16061740
- [Background] Atienza F, Almendral J, Moreno J, Vaidyanathan R, Talkachou A, Kalifa J, Arenal A, Villacastin JP, Torrecilla EG, Sanchez A, Ploutz-Snyder R, Jalife J, Berenfeld O. Activation of inward rectifier potassium channels accelerates atrial fibrillation in humans: evidence for a reentrant mechanism. Circulation. 2006 Dec 5;114(23):2434-42. doi: 10.1161/CIRCULATIONAHA.106.633735. Epub 2006 Nov 13. PMID 17101853
- [Background] Castells F, Mora C, Rieta JJ, Moratal-Perez D, Millet J. Estimation of atrial fibrillatory wave from single-lead atrial fibrillation electrocardiograms using principal component analysis concepts. Med Biol Eng Comput. 2005 Sep;43(5):557-60. doi: 10.1007/BF02351028. PMID 16411627
- [Background] Bollmann A, Sonne K, Esperer HD, Toepffer I, Klein HU. Patients with persistent atrial fibrillation taking oral verapamil exhibit a lower atrial frequency on the ECG. Ann Noninvasive Electrocardiol. 2002 Apr;7(2):92-7. doi: 10.1111/j.1542-474x.2002.tb00148.x. PMID 12049679
- [Background] Bollmann A, Binias KH, Toepffer I, Molling J, Geller C, Klein HU. Importance of left atrial diameter and atrial fibrillatory frequency for conversion of persistent atrial fibrillation with oral flecainide. Am J Cardiol. 2002 Nov 1;90(9):1011-4. doi: 10.1016/s0002-9149(02)02690-5. No abstract available. PMID 12398975
- [Background] Bollmann A, Kanuru NK, McTeague KK, Walter PF, DeLurgio DB, Langberg JJ. Frequency analysis of human atrial fibrillation using the surface electrocardiogram and its response to ibutilide. Am J Cardiol. 1998 Jun 15;81(12):1439-45. doi: 10.1016/s0002-9149(98)00210-0. PMID 9645894
- [Background] Burashnikov A, Di Diego JM, Zygmunt AC, Belardinelli L, Antzelevitch C. Atrium-selective sodium channel block as a strategy for suppression of atrial fibrillation: differences in sodium channel inactivation between atria and ventricles and the role of ranolazine. Circulation. 2007 Sep 25;116(13):1449-57. doi: 10.1161/CIRCULATIONAHA.107.704890. Epub 2007 Sep 4. PMID 17785620
- [Background] Fedida D, Orth PM, Chen JY, Lin S, Plouvier B, Jung G, Ezrin AM, Beatch GN. The mechanism of atrial antiarrhythmic action of RSD1235. J Cardiovasc Electrophysiol. 2005 Nov;16(11):1227-38. doi: 10.1111/j.1540-8167.2005.50028.x. PMID 16302909
- [Background] Duggan ST, Scott LJ. Intravenous vernakalant: a review of its use in the management of recent-onset atrial fibrillation. Drugs. 2011 Jan 22;71(2):237-52. doi: 10.2165/10489050-000000000-00000. PMID 21275448
- [Background] Feng J, Xu D, Wang Z, Nattel S. Ultrarapid delayed rectifier current inactivation in human atrial myocytes: properties and consequences. Am J Physiol. 1998 Nov;275(5):H1717-25. doi: 10.1152/ajpheart.1998.275.5.H1717. PMID 9815079
- [Background] Kneller J, Kalifa J, Zou R, Zaitsev AV, Warren M, Berenfeld O, Vigmond EJ, Leon LJ, Nattel S, Jalife J. Mechanisms of atrial fibrillation termination by pure sodium channel blockade in an ionically-realistic mathematical model. Circ Res. 2005 Mar 18;96(5):e35-47. doi: 10.1161/01.RES.0000160709.49633.2b. PMID 15731458
- [Background] Stiell IG, Roos JS, Kavanagh KM, Dickinson G. A multicenter, open-label study of vernakalant for the conversion of atrial fibrillation to sinus rhythm. Am Heart J. 2010 Jun;159(6):1095-101. doi: 10.1016/j.ahj.2010.02.035. PMID 20569725
- [Background] Yue L, Feng J, Gaspo R, Li GR, Wang Z, Nattel S. Ionic remodeling underlying action potential changes in a canine model of atrial fibrillation. Circ Res. 1997 Oct;81(4):512-25. doi: 10.1161/01.res.81.4.512. PMID 9314832
- [Background] Castells F, Cervigon R, Millet J. On the preprocessing of atrial electrograms in atrial fibrillation: understanding Botteron's approach. Pacing Clin Electrophysiol. 2014 Feb;37(2):133-43. doi: 10.1111/pace.12288. Epub 2013 Nov 12. PMID 24219142
- [Background] Castells F, Cebrian A, Millet J. The role of independent component analysis in the signal processing of ECG recordings. Biomed Tech (Berl). 2007 Feb;52(1):18-24. doi: 10.1515/BMT.2007.005. PMID 17313329
- [Background] Quintanilla JG, Moreno J, Archondo T, Chin A, Perez-Castellano N, Usandizaga E, Garcia-Torrent MJ, Molina-Morua R, Gonzalez P, Rodriguez-Bobada C, Macaya C, Perez-Villacastin J. KATP channel opening accelerates and stabilizes rotors in a swine heart model of ventricular fibrillation. Cardiovasc Res. 2013 Aug 1;99(3):576-85. doi: 10.1093/cvr/cvt093. Epub 2013 Apr 23. PMID 23612586
- [Background] Perez-Castellano N, Villacastin J, Salinas J, Vega M, Moreno J, Doblado M, Ruiz E, Macaya C. Epicardial connections between the pulmonary veins and left atrium: relevance for atrial fibrillation ablation. J Cardiovasc Electrophysiol. 2011 Feb;22(2):149-59. doi: 10.1111/j.1540-8167.2010.01873.x. Epub 2010 Aug 30. PMID 20807282
- [Background] Perez-Castellano N, Villacastin J, Aragoncillo P, Fantidis P, Sabate M, Garcia-Torrent MJ, Prieto C, Corral JM, Moreno J, Fernandez-Ortiz A, Vano E, Macaya C. Pathological effects of pulmonary vein beta-radiation in a swine model. J Cardiovasc Electrophysiol. 2006 Jun;17(6):662-9. doi: 10.1111/j.1540-8167.2006.00462.x. PMID 16836719